CLINICAL TRIAL: NCT01407679
Title: Efficacy and Safety of Oral Alitretinoin (Toctino®) in the Treatment of Patients With Cutaneous Lupus Erythematosus: A Multicentre, Open-Label, Prospective Pilot Study
Brief Title: Efficacy and Safety of Oral Alitretinoin (Toctino®) in the Treatment of Patients With Cutaneous Lupus Erythematosus
Acronym: AliCLE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKM 10_0019
Record Dates: First submitted 2011-08-01; First posted 2011-08-02 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Lupus Erythematosus, Cutaneous
Keywords: cutaneous lupus erythematosus; discoid lupus erythematosus; subacute cutaneous lupus erythematosus; lupus erythematosus tumidus
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Discoid | interventions — Alitretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alitretinoin (Experimental)
  Interventions: Drug: Alitretinoin

INTERVENTIONS:
Drug: Alitretinoin — 1 capsule Alitretinoin 30 mg per day; optional reduction to 10 mg per day in case unacceptable adverse reactions to the higher dose occur
  Other Names: Alitretinoin 30 mg soft capsules; Alitretinoin 10 mg soft capsules

SUMMARY:
To evaluate the therapeutic effect of oral alitretinoin (Toctino®) in the treatment of CLE with respect to proportion of responders based on the Revised Cutaneous Lupus Disease Area and Severity Index (RCLASI) activity score for skin lesions at baseline and after 24 weeks of treatment or at the latest assessment for patients who withdrew prematurely. Response is defined as a reduction of 50% in the total RCLASI compared to the baseline value ("RCLASI 50").

ELIGIBILITY:
Inclusion Criteria:

* A clinical and histological diagnosis of CLE (DLE, SCLE, LET) who failed to respond to topical corticosteroids;
* Total RCLASI activity score of skin lesions >6 (at least 3 points in at least 2 locations);
* At least one primary but preferably 2 methods of contraception;

Exclusion Criteria:

* Systemic Lupus Erythematosus (SLE) with major systemic organ involvement, e.g. clinical significant renal involvement, requiring systemic medical treatment for the disease;
* Clinically significant illness that may influence the outcome of the study in the four weeks before and during the study;
* Active severe infection diseases, including chronic or localized;
* Patients with hepatic insufficiency (AST, ALT > 2.5 x ULN), severe renal failure (creatinine clearance < 60ml/min), or hypercholesterolemia characterized by:

  1. Fasting triglyceridemia > 1.5 x upper limit of normal (ULN)
  2. Fasting total cholesterol > 1.5 x ULN
  3. Fasting low-density lipoprotein (LDL) cholesterol > 1.5x ULN
* Patients with known hypersensitivity to other retinoids or vitamin A derivatives, or to any study medication component, especially soybean oil and partly hydrogenated soybean oil;
* Patients with cardiovascular risk factors that would exclude a starting dose of 30 mg of alitretinoin;
* Topical corticosteroids within 14 days prior to dosing;
* Patients treated with any systemic or topical retinoids within 4 weeks before start of study treatment;
* Drugs with a potential for drug-drug interaction, such as systemic tetracyclines, ketoconazole, or St. John"s Wort within 1 week, or receiving systemic itraconazole within 2 weeks, before start of study treatment;
* Initiation or change in the dose of any current systemic medication for the treatment of CLE/SLE prior to the study (time depending on drug class and half-life);
* Treatment with immunosuppressive drugs for other reasons, 4 weeks prior and within the study;
* Concomitant medication with drugs with a known photosensitizing potential, e.g. tetracyclines, griseofulvin, thiazides, furosemide, sulfonamides or tolbutamide;
* Drugs associated to CLE-induction: terbinafine, hydrochlorothiazide, diltiazem, verapamil, nifedipine, nitrendipine, fluorouracil, penicillamine, infliximab, adalimumab, etanercept, pantoprazole;

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Primary efficacy outcome is the response rate at week 24 or at the latest assessment for patients who withdrew prematurely. | Week 24 or at the latest assessment for patients who withdrew prematurely.
  Response is defined as a reduction of 50% in the total RCLASI activity for skin lesions, compared to the baseline value ("RCLASI 50")

SECONDARY OUTCOMES:
Proportion of patients with RCLASI 50 at week 12 of treatment. | Week 12 of treatment
Proportion of patients with at least partial response at end of therapy (with regard to RCLASI activity score for skin lesions). | End of therapy (up to 24 weeks)
Patient's global assessment and VAS for itch and pain 12 weeks after the beginning of treatment. | 12 weeks after the beginning of treatment
Number of Participants with Adverse Events (AEs) and their severity. | 24 weeks of treatment + 5 weeks of follow up
Patient's global assessment and VAS for itch and pain at the end of therapy. | End of therapy (up to 24 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Kuhn, Prof. Dr., Principal Investigator — Department of Dermatology, University Hospital Muenster, Muenster, Germany
Locations (3):
- Germany (3):
  - Department of Dematology, University Hospital, Mannheim, Baden-Wurttemberg
  - Department of Dermatology, Ludwig-Maximilians University, Munich, Bavaria
  - Department of Dermatology, University Hospital, Münster, Westfalen